CLINICAL TRIAL: NCT05419466
Title: Kinetic of Plasmatic Compounds and Metabolites of a Melatonin-based Formulation in Healthy Subjects
Brief Title: Kinetic of Compounds of a Melatonin-based Formulation in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Larena SAS (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C1711
Record Dates: First submitted 2022-06-03; First posted 2022-06-15 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Melatonin Bioavailability
MeSH Terms: interventions — Dietary Supplements; Zinc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- melatonin and zinc bioavailability (Experimental): dietary supplement, 1 tablet containing delayed release melatonin, zinc and lemon balm
  Interventions: Dietary Supplement: dietary supplement, 1 tablet containing delayed release melatonin, zinc and lemon balm

INTERVENTIONS:
Dietary Supplement: dietary supplement, 1 tablet containing delayed release melatonin, zinc and lemon balm — dietary supplement is dosed at 1.9 mg of melatonin, 10 mg of zinc and 200 mg of lemon balm for one tablet

SUMMARY:
This study is conducted to clinically document the melatonin and zinc bioavailability of a dietary supplement containing delayed release melatonin, zinc and lemon balm

ELIGIBILITY:
Inclusion Criteria:

* Male between the ages of 18 and 45,
* In good general health, i.e., free of chronic conditions and not taking medication at the time of inclusion and/or long-term,
* Over 70 kg and with a body mass index between 18.5 and 24.9,
* Able and willing to participate in the research by complying with the procedures of the protocol, in particular concerning the taking of the product under study and the performance of sequential blood tests,
* Having freely signed the consent form after adequate information on the proposed study,
* Affiliated to a social security scheme or similar.

Exclusion Criteria:

* Smoker,
* Drug addict,
* Subject with an alcohol consumption of more than 2 glasses per day,
* Taking a drug treatment or melatonin or zinc or a product containing it within 48 hours prior to a kinetics visit,
* Known organic or functional abnormality of the urinary tree,
* Any medical condition that would involve a change in melatonin metabolism: Drug intake: Fluvoxamine, 5- or 8-methoxypsoralen, cimetidine, carbamazepine, rifampicin, analgesics, Liver abnormality known or detected at the screening visit and judged to be clinically significant by the investigator, Known autoimmune disease,
* Any condition that could involve zinc deficiency or hyperzincemia: Medication intake: penicillamine or diuretics, Poisoning by exposure to zinc (zinc mines, zinc metallurgy, galvanizing operations, manufacture of alloys, use of zinc-based pigments and salts, etc.), Pick's disease, malabsorption (pancreatic insufficiency, biliary obstruction, gastrectomy, jejuno-ileostomy, intestinal diverticulum, tropical sprue, celiac disease, cystic fibrosis), intestinal inflammation (enteropathy with protein leakage, inflammatory colitis), liver disorders (cirrhosis, hepatitis) , kidney disorders (chronic renal failure, nephrotic syndrome), neuropsychiatric disorders (anorexia nervosa, endogenous depression, alcoholism), genetic diseases (acrodermatitis enteropathica, thalassemia, sickle cell disease, diabetes, trisomy 21, phenylketonuria), parasitic diseases (ankylostomiasis, schistosomiasis, malaria , giardiasis)
* Subject assessed as "rather" or "definitely" among evening people,
* Epileptic subject,
* Asthmatic subject,
* Known hypertension (>140/90),
* Diagnosis of migraine by a health professional according to the International Headache Society (IHS) criteria revised in 2004,
* With a sleep disorder,
* Thyroid dysfunction, hyperglycemia or anemia judged to be clinically significant by the investigator,
* Blood donation within one month prior to inclusion,
* A known organic or psychological abnormality (including a history of severe depression) that may bias the results of the study as judged by the investigator,
* Workers with atypical working hours (night work, staggered working hours),
* Known allergy or intolerance to any of the components of the product,
* Psychological or linguistic inability to understand and sign informed consent,
* Participant in another interventional clinical trial or during a period of exclusion from a previous clinical trial,
* Under legal protection (guardianship, curatorship) or deprived of his rights as a result of the administrative or judicial decision,
* Subject who has reached the maximum threshold for compensation for research provided for in the regulations.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-03-14 (Actual); Primary Completion 2023-05-22 (Actual); Study Completion 2023-05-22 (Actual)

PRIMARY OUTCOMES:
Evolution of the plasma melatonin concentration | Up to 720 minutes after taking the tablet
  The change in plasma melatonin concentration

SECONDARY OUTCOMES:
Plasma melatonin AUC | Up to 720 minutes after taking the tablet
  Area Under the Curve of plasma melatonin
Plasma melatonin Cmax | Up to 720 minutes after taking the tablet
  Peak concentration of plasma melatonin
Plasma melatonin Tmax | Up to 720 minutes after taking the tablet
  Time take to reach Cmax of plasma melatonin
Plasma melatonin half life | Up to 720 minutes after taking the tablet
  Time required for the concentration of plasma melatonin to decrease to half of its starting dose
Evolution of the plasma concentration of 6-sulfatoxymelatonin | Up to 720 minutes after taking the tablet
  The change in plasma 6-sulfatoxymelatonin concentration
Plasma 6-sulfatoxymelatonin AUC | Up to 720 minutes after taking the tablet
  Area Under the Curve of plasma 6-sulfatoxymelatonin
Plasma 6-sulfatoxymelatonin Cmax | Up to 720 minutes after taking the tablet
  Peak concentration of plasma 6-sulfatoxymelatonin
Plasma 6-sulfatoxymelatonin Tmax | Up to 720 minutes after taking the tablet
  Time take to reach Cmax of plasma 6-sulfatoxymelatonin
Plasma 6-sulfatoxymelatonin half life | Up to 720 minutes after taking the tablet
  Time required for the concentration of plasma 6-sulfatoxymelatonin to decrease to half of its starting dose
Evolution of the plasma zinc concentration | Up to 720 minutes after taking the tablet
  The change in plasma zinc concentration
Plasma zinc AUC | Up to 720 minutes after taking the tablet
  Area Under the Curve of plasma zinc
Plasma zinc Cmax | Up to 720 minutes after taking the tablet
  Peak concentration of plasma zinc
Plasma zinc Tmax | Up to 720 minutes after taking the tablet
  Time take to reach Cmax of plasma zinc
Plasma zinc half life | Up to 720 minutes after taking the tablet
  Time required for the concentration of plasma zinc to decrease to half of its starting dose
Evolution of state of drowsiness | Up to 720 minutes after taking the tablet
  The change in (Visual Analog Scale)VAS score, minimum = 0 and maximum = 10 higher score means a worse outcome
Adverse events | During study participation, maximum 45 days
  Number and type of adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Claustrat, Study Director — PiLeJe
Locations (1):
- Cen Experimental, Dijon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ait Abdellah S, Gal C, Guinobert I, Bardot V, Raverot V, Vitacca A, Blondeau C, Claustrat B. Melatonin Bioavailability After Oral Administration of a New Delayed-Release Form in Healthy Male Volunteers. Drugs R D. 2024 Sep;24(3):415-423. doi: 10.1007/s40268-024-00482-6. Epub 2024 Aug 22. PMID 39174857